CLINICAL TRIAL: NCT05889754
Title: The Validity and Reliability of the Turkish Version of the "Pediatric Haemophilia Activities List - Short - PedHALshort" Questionnaire
Brief Title: Reliability and Validity of the Turkish Version of the PedHAL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Tuğba GÖNEN, Assistant Professor, Hasan Kalyoncu University
Other Study IDs: 2023/53
Record Dates: First submitted 2023-05-22; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Hemophilia; Hemophilia A, Severe; Hemophilia B
Keywords: Functional independence; Activities of daily living; Hemophilia; Factor VIII; Factor IX
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemophilia Group: The PedHAL questionnaire will be administered to children aged 4-17 years with a diagnosis of hemophilia twice, one week apart. For construct validity assessment, the questionnaire will be compared with the Hemophilia Functional Independence Score (HJHS).

SUMMARY:
This study aimed to establish the validity and reliability of the Turkish version of the Pediatric Haemophilia Activities List (short - PedHALshort) questionnaire.

DETAILED DESCRIPTION:
Hemophilia is a blood disease characterized by a bleeding disorder that develops due to the deficiency of clotting factor VIII (Hamophilia A) or coagulation factor IX (Hamophilia B) proteins that provide clotting in the blood. In the hereditary disease showing X-linked recessive inheritance, female individuals are carriers and male individuals show a clinical picture. Although the clinical picture changes depending on the duration and frequency of bleeding, the severity of the disease is classified as severe, moderate and mild. Musculoskeletal problems are the most common complications in patients with severe and moderate hemophilia. Hemarthroses due to bleeding in the joint (80%) and hematomas due to intramuscular bleeding (20%) cause joint degeneration and muscle atrophy. Recurrent hemarthroses occur when there is not enough clotting factor in the setting, often before the previous hemarthrosis has resolved. This creates a vicious cycle of bleeding-inflammation-rebleeding known as the "target joint". The resulting vicious circle causes permanent damage to bone and cartilage structures and causes "arthropathy". The knee is the joint region where hemarthrosis and arthropathy are most common, followed by the elbow and ankle joints. Since these joints in the musculoskeletal system contain more synovial tissue than the others, they are more exposed to trauma and load and are injured. As a result of all these, pain, joint limitations and muscle strength losses occur. All these clinical findings lead to a decrease in functional independence in activities of daily living with the restriction of physical activity in patients.

In the literature, there are questionnaires and measurement methods in which many functional evaluations are made for hemophilia patients. However, most of them have not been validated and reliable in Turkish. For this purpose, our study aimed to establish the validity and reliability of the Turkish version of the Pediatric Haemophilia Activities List (PedHALshort) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Hemophilia by a physician (Factor VIII-IX)
* Ages 4-17 years old
* Receiving regular prophylactic treatment
* Children who volunteered to participate in the study and whose family consent was given

Exclusion Criteria:

- Children with neurological signs that limit activities of daily living

Ages: 4 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Hemophilia a disease is an X-linked recessive disease. Therefore, girls become carriers and do not show muscle joint problems.
Study Population: Pediatric group hemophilia A and hemophilia B children living in Gaziantep constitute the study population.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-30 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Paediatric Haemophilia Activities List | through of the study, average 6 months
  PedHAL contains 22 items in 7 areas: sitting/kneeling/standing, functions of legs, functions of arms, use of transportation, personal care, housework and leisure activities, and sports. It consists of a child version (8-17 years old) and a parent version (4-17 years old). Items are scored for each item on a 6-point Likert scale ("impossible", "always", "usually", "sometimes", "almost never", "never"), "not applicable (N/A)". . The score is converted to a normalized score from 0 to 100, the higher score representing better functional status. If more than half of the items are missing or scored as "not applicable" (N/A), a valid total score will not be calculated.
FISH | through of the study, average 6 months
  The scoring system, which is categorized according to the international classification of functionality, disability and health (ICF), has been prepared by considering the activities that hemophilia patients may be affected by in their daily lives. Being a performance-based scale allows it to be used in different languages. The scale consists of 8 questions in total, including the sub-parameters of self-care, transfer and locomotion. Self care subparameter; eating-hygiene, bathing and dressing, transfer sub-parameter; chair and squat, locomotion subparameter; It consists of walking, stair climbing (12-14 steps) and running activities.
  Scoring of the activities is between 1 and 4 according to the degree of independence. The minimum score that can be obtained from the scale is 8, and the maximum score is 32. A high score indicates the functional independence of the individual.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Souza JC, Simoes HG, Campbell CS, Pontes FL, Boullosa DA, Prestes J. Haemophilia and exercise. Int J Sports Med. 2012 Feb;33(2):83-8. doi: 10.1055/s-0031-1286292. Epub 2011 Nov 17. PMID 22095329
- [Background] Wagner B, Kruger S, Hilberg T, Ay C, Hasenoehrl T, Huber DF, Crevenna R. The effect of resistance exercise on strength and safety outcome for people with haemophilia: A systematic review. Haemophilia. 2020 Mar;26(2):200-215. doi: 10.1111/hae.13938. Epub 2020 Feb 24. PMID 32091659
- [Background] Schafer GS, Valderramas S, Gomes AR, Budib MB, Wolff AL, Ramos AA. Physical exercise, pain and musculoskeletal function in patients with haemophilia: a systematic review. Haemophilia. 2016 May;22(3):e119-29. doi: 10.1111/hae.12909. Epub 2016 Apr 14. PMID 27075748
- [Background] De la Corte-Rodriguez H, Rodriguez-Merchan EC. The role of physical medicine and rehabilitation in haemophiliac patients. Blood Coagul Fibrinolysis. 2013 Jan;24(1):1-9. doi: 10.1097/MBC.0b013e32835a72f3. PMID 23103725
- [Background] Young NL, Bradley CS, Blanchette V, Wakefield CD, Barnard D, Wu JK, McCusker PJ. Development of a health-related quality of life measure for boys with haemophilia: the Canadian Haemophilia Outcomes--Kids Life Assessment Tool (CHO-KLAT). Haemophilia. 2004 Mar;10 Suppl 1:34-43. doi: 10.1111/j.1355-0691.2004.00877.x. PMID 14987247
- [Background] Timmer MA, Gouw SC, Feldman BM, Zwagemaker A, de Kleijn P, Pisters MF, Schutgens REG, Blanchette V, Srivastava A, David JA, Fischer K, van der Net J. Measuring activities and participation in persons with haemophilia: A systematic review of commonly used instruments. Haemophilia. 2018 Mar;24(2):e33-e49. doi: 10.1111/hae.13367. Epub 2017 Nov 27. PMID 29178149
- [Background] Shrout PE, Fleiss JL. Intraclass correlations: uses in assessing rater reliability. Psychol Bull. 1979 Mar;86(2):420-8. doi: 10.1037//0033-2909.86.2.420. PMID 18839484